CLINICAL TRIAL: NCT04662736
Title: Tedizolid Suppressive Antimicrobial Therapy
Brief Title: Tedizolid Suppressive Antimicrobial Therapy in a Reference Center
Acronym: TediSAT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 232
Record Dates: First submitted 2020-11-25; First posted 2020-12-10 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Bone and Joint Infection
Keywords: bone and joint infection; tedizolid; suppressive antibiotic therapy
MeSH Terms: interventions — tedizolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had a BJI/PJI treated with tedizolid as a suppressive antibiotic therapy
  Interventions: Other: patients having had a BJI/PJI treated with tedizolid as a suppressive antibiotic therapy

INTERVENTIONS:
Other: patients having had a BJI/PJI treated with tedizolid as a suppressive antibiotic therapy — description of osteo-articular infection managed with tedizolid as a suppressive antibiotic therapy

SUMMARY:
the aim of the study is to describe the management and outcome of patients having an osteo-articular infection treated by tedizolid as a suppressive antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients having an osteo-articular infection treated with tedizolid as a suppressive antibiotic therapy

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients having an osteo-articular infection treated with tedizolid as a suppressive antibiotic therapy managed at the CRIOAc LYON, Croix-Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
rate of patients having had a BJI/PJI treated with tedizolid as a suppressive antibiotic therapy | between 2016 and 2021
  proportion of patients having tedizolid as a suppressive antibiotic therapy
rate of failure in patients having had a BJI/PJI treated with tedizolid as a suppressive antibiotic | 2 years
  proportion of patients having a failure under tedizolid as a suppressive antibiotic therapy
rate of adverse event in patients having had a BJI/PJI treated with tedizolid as a suppressive | through study completion, an average of 1 year
  proportion of patients having a adverse event under tedizolid as a suppressive antibiotic therapy
Description of patients having had a BJI/PJI treated with tedizolid as a suppressive | 2 years
  type of patients: age, CMI, comorbidities...
Description of BJI/PJI treated with tedizolid as a suppressive | 2 years
  implant or prothese or not, acute/ chronic, bacteriology

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/